CLINICAL TRIAL: NCT05136859
Title: Inflammatory Marker and Pre-existing Venous Fibrosis to Predict AVF Mal-maturation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202006195RINC
Record Dates: First submitted 2021-11-10; First posted 2021-11-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Arteriovenous Fistula
Keywords: hemodialysis; Inflammation; Arteriovenous Fistula; perivascular fat
MeSH Terms: conditions — Arteriovenous Fistula; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preserve (Experimental): preserve the perivascular fat of the target cephalic vein
  Interventions: Procedure: preserve
- remove (No Intervention): remove from perivascular fat of the target cephalic vein

INTERVENTIONS:
Procedure: preserve — preserve the perivascular fat of the target cephalic vein
  Arms: preserve

SUMMARY:
End-stage renal disease patients needs a functional vascular access to receive hemodialysis and prolong their lives. Arteriovenous fistula (AVF) is priority consideration for hemodialysis, which is a connecting a superficial vein to a nearby artery and allowing this vein to enlarge and increase in internal diameter under arterial circulation. Unfortunately, 30-50% of fistulae fail to mature. Vascular calcification and stenosis were considered for early failure. The perivascular fat of artery can be predicted successful AVF maturation. However, Few previous studies have compared AVF maturation between perivascular the fat of cephalic vein or removal during the AVF surgery. This study evaluated whether the effect of AVF inflammation and preexisting vascular fibrosis is associated to perivascular the fat of cephalic vein. Investigators will also verify inflammation by analysis of blood and tissue samples, the association of pre-existing fibrosis, and the clinical correlation with AVF early failure.

This study will enroll patients with chronic kidney disease stage 5 and stage 6 who will need maintenance-hemodialysis (HD) from Nov 2021 to Dec 2022. Investigators will use the preoperative ultrasound assessment tool to confirm the feasibility of the arm vessels for the creation of a native AVF. As a prospective randomized controlled trial of perivascular fat preservation or removal during the AVF surgery, a study assistant will help the randomization and explain the informed consent to the patient . The subjects are randomly split into two groups: the experimental group will have the perivascular fat of the target cephalic vein preserved the control group will have the fat removed before the AVF anastomosis. The survey will enroll 100 adult patients and categorize them into groups according to each AVF maturation, JAS, or FTM (see definition below) by 3 - 12 after the surgery.

DETAILED DESCRIPTION:
The arteriovenous fistula (AVF) is the preferred vascular access for hemodialysis, which is surgically created but connecting a superficial vein to nearby artery and allowing this vein to enlarge and increase in internal diameter under arterial circulation. Successful fistula maturation depends on dilatation and remodeling of the artery and vein, but the stiff and thickened vessels of end-stage renal diseases (ESRD) patients may respond poorly to signals that promote these adaptations. About 20 - 40% of AVFs maturation fails and no effective treatment to prevent AVF maturation failure. Paulson WD summarized four points for maturation failure. Surgical skill; preexisting vascular disease; Upstream events; and Downstream events. Upstream events are the mechanisms that initially cause injury to the endothelium (surgical trauma, hemodynamic shear stress, vessel wall injury caused by needle punctures, etc.). Downstream events are the responses to endothelial injury (leukocyte adhesion, migration of smooth muscle cells from the media to the intimal layer, smooth muscle proliferation, etc.). However, upstream and downstream events are important steps in maturation failure, preexisting vascular disease should not be neglected as it sets the stage for what follows. Medial collagen fibers are organized into lamellar units and oriented circumferentially with crimps in healthy blood vessels. However, higher medial collagen content maybe stiffer and limited ability to dilate. Recently, researches have shows preexisting fibrosis condition in veins was associated with maturation.

Inflammation for AVF setting can be divided into two parts: local and systemic inflammation. For local inflammation had been indicated caused by the trauma of fistula creation and local hypoxia; For systemic inflammation, which occurs because of uremia present in CKD patients. Recent study have suggested AVF failure was linked to inflammation. The perivascular fat of artery can be predicted successful AVF maturation. Lipectomy of cephalic vein is a routine method during hemodialysis arteriovenous fistula creation[9]. However, Few previous studies have compared AVF maturation between perivascular the fat of cephalic vein or removal during the AVF surgery.

Specific aims

Successful fistula maturation depends upon dilatation and remodeling of the artery and vein, but the stiff and thickened vessels of ESRD patients may respond poorly to signals that promote these adaptations. Although our preliminary data showed that preexisting vascular fibrosis increased in AVFs failure. But the finding still needs more verifications. In this study, Investigators will focus on the finding of molecular marks to be related to AVFs maturation or failure. The study include the following sections:

1. Whether vascular fibrosis exists in AVF patients and its association with maturation failure.
2. Whether vascular fibrosis is associated with inflammation.
3. Examine the cytokines expression of neutrophil in blood.
4. Whether the perivascular fat of cephalic vein is associated with AVF failure

Aim 1. Whether vascular fibrosis exists in AVF patients and its association with maturation failure. Investigators will observe vascular fibrosis by histopathology and western blot.

First of all, the subjects are those adult uremic patients who will undergo an AVF creation. The survey will enroll the patients with chronic kidney disease (CKD) stage 5 (CKD-5) and stage 6 (CKD-6) who will need maintenance-hemodialysis (HD). Investigators will use the preoperative ultrasound assessment tool to confirm the feasibility of the arm vessels for the creation of a native AVF.

As a prospective randomized controlled trial of perivascular fat preservation or removal during the AVF surgery, a study assistant will help the randomization and explain the informed consent to the patient. The subjects are randomly split into two groups: the experimental group will have the perivascular fat of the target cephalic vein preserved the control group will have the fat removed before the AVF anastomosis.

The surgeon will harvest the distal vein stump and 1 cm of subcutaneous fat for at least 1.5-cm in length during an AVF creation, at the same time will get a 10-cc plasma sample. The survey will enroll 100 adult patients and categorize them into groups according to each AVF maturation, JAS, or FTM (see definition below) by 3 - 12 after the surgery.

Preoperative vascular ultrasound assessment.

All patients will have clinical and ultrasound exam to assess the suitability of surgery, The patient will be excluded If their vessels and/or clinical condition are not suitable used to hemodialysis. A hemodialysis arteriovenous fistula (HDAVF) maturity score based on the following three objective ultrasonic measurements. Give a summary score range from 0 to 9 points. Higher scores indicating more mature. Ultrasound testing parameters are defined as follows:

1. Measuring the arm artery diameter and total blood flow. The brachial artery is defined as measured from the proximal 4 (+/- 2,2 to 6) cms within the curved line of the elbow, Investigators will measure the vascular diameter and estimate total forearm blood flow.
2. Radial artery scan of the forearm is defined as the diameter of the radial artery scanned from the start of the antecubital to the wrist.line. Notedly, Investigators also confirm its diameter> = 2.0 mm and identify no obvious stenosis of the antecubital to the wrist.line. Notedly, Investigators also confirm its diameter> = 2.0 mm and identify no obvious stenosis.
3. Measure the non-augmented diameter of the cephalic vein. The midpoint of it is defined as the middle between the elbow line and the wrist line, Which is around 10 (+/- 2, 8 ~ 12) cms distal to the elbow.
4. Measure the augmented diameter of the cephalic vein. Pressure is applied to the upper arm with tourniquet cuff to 100-mm-Hg temporarily and which provides moderate resistance, wait 30 seconds, then investigators measure the cephalic vein where has been defined above. Accordingly, the definition of venous compliance is defined as the degree of venous dilatation of the cephalic vein before and after augmentation. Furthermore, the compliance of vein is defined as the percentage of augmented / non-augmented cross-section area of the vein.
5. Investigators will confirm the whole segment of cephalic vein is to be> 2.0 mm in diameter and identify no significant stenosis.

Definition of clinical success: It is defined as the target HDAVF can be used by two needles and complete the HD session for at least ⅔ of prescribing sessions in a month. A minimum criterion of a run is at an average blood flow rate of 300 ml/min in a 3.5-hour HD session to achieve a target sp-Kt/V of 1.2.14 In which a successful HD session is defined as completion of HD with a dialysis flow rate is more than 200 ml/min, and a session duration of 4 hours or more.

Definition of success by ultrasound parameters: the survey proposes an objective ultrasound scoring system and considers a total score of four or more as AVF maturation.

For histology analysis, samples were paraffin-embedded and sectioned. H&E (hematoxylin and eosin) are common stains used in histology. The hematoxylin stains cell nuclei is blue, and eosin stains the extracellular matrix and cytoplasm presents pink. The Movat pentachrome staining can be demonstrated that collagen, elastin, muscle mucin and fibrin in tissue sections. Investigators use Sirius-red staining to observe the collagen I and III fibers in tissue sections. In order to detect calcium deposits, Investigators use Alizan red staining. The Masson's trichrome will be used to stain. In the trichrome stain, smooth muscle appears red, and collagen appears blue.

For western blot assay, collagen, α-SMA, TIMP-1, and TIMP2 expression will increase in vascular fibrosis. Hence, investigators will detect expression of collagen, α-SMA, MMP-9, MMP2, TIMP-1, TIMP2 in AVF maturation and failure tissue. Tissues were homogenized and lysed. Protein concentration for each tissue extract was determined using a BCA protein assay according to the instructions of the supplier (Pierce Chemical Co., Rockford, Illinois, USA). Fifty microgram of tissue lysates protein per lane were separated by SDS-PAGE under reducing conditions and blotted onto PVDF membranes (Millipore Corp., Bedford, Massachusetts, USA). Membranes were blocked in 5% defatted dry milk/ PBS/0.1% Tween-20 (PBST) and were then incubated with the primary antibody for 1 hour. Blots were washed 4 times PBST, and the secondary peroxidase-conjugated antibody (Jackson ImmunoResearch Labora-tories Inc., West Grove, Pennsylvania, USA) was added (1:10,000) for another hour. Finally, membranes were washed in PBST, and detection of the antigen was carried out using the enhanced chemiluminescence detection method according to the manufacturer's recommendations

Aim 2. Whether vascular fibrosis is associated with inflammation. Inflammation in the setting of AVF was involved locally and systemically. Local inflammation caused by trauma of fistula creation and local hypoxia. So, investigators will measure the IL8, IL1b, IL6, IL10, TNF, IL12p70, CCL5(RANTES), CXCL9 (MIG), CCL2 (MCP1), IP10 and compare expression between AVF maturation and failure tissue by QPCR and Multiplex ELISA. Beside, systemic inflammation occurs because of uremia that is present in chronic kidney diseases. Also, investigators will detect expression of IL8, IL1b, IL6, IL10, TNF, IL12p70, CCL5(RANTES), CXCL9 (MIG), CCL2 (MCP1), IP10 and compare expression between AVF maturation and failure serum by CBA assay.

For QPCR assay, RNA was extracted from vein tissue by the TRIzol protocol (Life Technologies, Invitrogen). RNA concentrations were quantified by Nanodrop. The purity of the total RNA extracted was determined as the 260/280 nm ratio and the integrity was checked. QPCR was performed by the TaqMan system.

For ELISA assay, tissues were lysed in PBS buffer and using commercial ELISA kits (R&D) according to the manufacturer's protocol. The lysates were normalized to the total protein content determined using a commercial BCA protein assay kit.

For Cytokine Bead Array (CBA) assay, the Human Inflammatory Cytokines CBA Kit (BD Biosciences, San Jose, CA) was used, which measures all of the above cytokines except GM-CSF, IL-2, and IFN-γ; data were acquired on a BDTM FACS caliber flow cytometer. Both assays were performed according to the manufacturer's instructions except for the use of modified calibration curves as described below. All standards and samples were measured in duplicate.

Aim 3. Examine the cytokines expression profile of neutrophilic in blood. To perform this, investigators will examine the peripheral blood neutrophil population by flow cytometry stain with CD11b+/CD66b/CD34/CD45. Next to determine the percentage of neutrophils expressing target cytokines in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20 and older adult patients.
2. preoperatively clinical and ultrasound assessment of the arm vessels are visible for the creation of a native HDAVF that include：the augmented diameters of the veins is > 2.0 mm and the diameter of the radial artery is> 2.0 mm. Besides, there is no obvious stenosis of vessels in the forearm.

Exclusion Criteria:

1. The patient refused to join the study
2. serious heart failure (Physicians identify insufficient cardiac output that may affect sacral blood flow development after surgery)
3. Unconsciousness
4. Bedridden for long time
5. systemic lupus erythematosus(SLE), or other known autoimmune diseases
6. The physician excludes the possibility of creating a wrist HDAVF before surgery
7. Surgeon preoperatively identifies vessel inadequacy for the creation of a wrist HDAVF
8. Choose a site other than the wrist for surgery
9. Unexpected complications happen during the surgery that prevent the completion of a wrist HDAVF

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The success by ultrasound parameters. | 3 months after surgery
  Investigators propose an objective ultrasound scoring system(A hemodialysis arteriovenous fistula maturity score based on the following three objective ultrasonic measurements). Higher scores indicating more mature. Give a summary score range from 0 to 9 points., and of which a total of score 4 or more is considered as HDAVF maturation.
Definition of delay maturation | 3 months after surgery
  The subject HDAVF is clinically un-feasible for use for HD within 3 months and/or the A hemodialysis arteriovenous fistula maturity score(AFMS) based on the following three objective ultrasonic measurements(0-9) is less than 4.
  within 3 months and/or the A hemodialysis arteriovenous fistula maturity score based on the following three objective ultrasonic measurements is less than 4(AVF maturity score based on the following three objective ultrasonic measurements. 0 to 9.).

SECONDARY OUTCOMES:
The subject HDAVF is clinically un-feasible for use for HD within 3 months and/or the A hemodialysis arteriovenous fistula maturity score(AFMS) based on the following three objective ultrasonic measurements(0-9) is less than 4. | 3 months after surgery
  infection, bleeding, stroke, MI, deep vein thrombosis,peripheral arterial occlusion disease, died

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Martinez L, Duque JC, Tabbara M, Paez A, Selman G, Hernandez DR, Sundberg CA, Tey JCS, Shiu YT, Cheung AK, Allon M, Velazquez OC, Salman LH, Vazquez-Padron RI. Fibrotic Venous Remodeling and Nonmaturation of Arteriovenous Fistulas. J Am Soc Nephrol. 2018 Mar;29(3):1030-1040. doi: 10.1681/ASN.2017050559. Epub 2018 Jan 2. PMID 29295872
- [Result] Kheda MF, Brenner LE, Patel MJ, Wynn JJ, White JJ, Prisant LM, Jones SA, Paulson WD. Influence of arterial elasticity and vessel dilatation on arteriovenous fistula maturation: a prospective cohort study. Nephrol Dial Transplant. 2010 Feb;25(2):525-31. doi: 10.1093/ndt/gfp462. Epub 2009 Sep 15. PMID 19755475
- [Result] Holzapfel GA. Collagen in arterial walls: biomechanical aspects. In: Collagen. Springer; 2008:285-324.
- [Result] Shiu YT, Litovsky SH, Cheung AK, Pike DB, Tey JCS, Zhang Y, Young CJ, Robbin M, Hoyt K, Allon M. Preoperative Vascular Medial Fibrosis and Arteriovenous Fistula Development. Clin J Am Soc Nephrol. 2016 Sep 7;11(9):1615-1623. doi: 10.2215/CJN.00500116. Epub 2016 Aug 30. PMID 27577243
- [Result] Brahmbhatt A, Remuzzi A, Franzoni M, Misra S. The molecular mechanisms of hemodialysis vascular access failure. Kidney Int. 2016 Feb;89(2):303-316. doi: 10.1016/j.kint.2015.12.019. PMID 26806833
- [Result] Lee HS, Park MJ, Yoon SY, Joo N, Song YR, Kim HJ, Kim SG, Nizet V, Kim JK. Role of peribrachial fat as a key determinant of brachial artery dilatation for successful arteriovenous fistula maturation in hemodialysis patients. Sci Rep. 2020 Mar 2;10(1):3841. doi: 10.1038/s41598-020-60734-8. PMID 32123226
- [Result] Bourquelot P, Tawakol JB, Gaudric J, Natario A, Franco G, Turmel-Rodrigues L, Van Laere O, Raynaud A. Lipectomy as a new approach to secondary procedure superficialization of direct autogenous forearm radial-cephalic arteriovenous accesses for hemodialysis. J Vasc Surg. 2009 Aug;50(2):369-74, 374.e1. doi: 10.1016/j.jvs.2009.03.009. PMID 19631871
- [Result] Lee T, Mokrzycki M, Moist L, Maya I, Vazquez M, Lok CE; North American Vascular Access Consortium. Standardized definitions for hemodialysis vascular access. Semin Dial. 2011 Sep-Oct;24(5):515-24. doi: 10.1111/j.1525-139X.2011.00969.x. Epub 2011 Sep 9. PMID 21906166
- [Result] Murphy EA, Ross RA, Jones RG, Gandy SJ, Aristokleous N, Salsano M, Weir-McCall JR, Matthew S, Houston JG. Imaging in Vascular Access. Cardiovasc Eng Technol. 2017 Sep;8(3):255-272. doi: 10.1007/s13239-017-0317-y. Epub 2017 Jul 13. PMID 28707187